CLINICAL TRIAL: NCT01065545
Title: A Phase I Feasibility Study Assessing the Role of Maintenance Oral Clofarabine in Older Adults With Acute Myeloid Leukemia
Brief Title: The Role of Maintenance Oral Clofarabine in Older Adults With Acute Myeloid Leukemia
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to funding issues.
Sponsor: Northwestern University (Other)
Collaborators: Loyola University (Other); Rush University Medical Center (Other); University of Illinois at Chicago (Other); Genzyme, a Sanofi Company (Industry)
Responsible Party: Jessica Altman, MD, Northwestern University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 08H6; STU00008055 (Other: Northwestern University IRB)
Record Dates: First submitted 2010-02-08; First posted 2010-02-09 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Acute Myeloid Leukemia
Keywords: leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia | interventions — Clofarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Clofarabine (Experimental)
  Interventions: Drug: Clofarabine

INTERVENTIONS:
Drug: Clofarabine — dose escalation, administered orally, once a day for 21 days per cycle (cycles begin every 28-49 days)
  Other Names: CLOLAR; CAFda; Cl-F-ara-A

SUMMARY:
The purpose of this study is to determine the side effects of the study drug, clofarabine, when given by mouth to patients with acute myeloid leukemia (AML), in remission.

DETAILED DESCRIPTION:
Standard induction chemotherapy (chemotherapy given with the intent of inducing a remission/disappearance of the cancer) can lead to a complete remission (CR) in a large percentage (60% to 80%) of younger patients with newly diagnosed AML. However, the majority of patients relapse (their disease returns) despite intensive consolidation chemotherapy. In most chemotherapy studies, only a small percentage (30% to 40%) of patients who achieve a CR still are disease-free 5 years later. The outcome for older adults is even less favorable. Approximately 75% of elderly patients who achieve CR will relapse after 2 years or less and the toxicities seen with treatment are significant. A number of studies have shown that chemotherapy given to older adults after a remission has not improved this outcome; therefore new treatments need to be investigated. Clofarabine is a drug that has been studied in older adults who have achieved a CR. The treatment was found to have fewer side effects then other consolidation therapies. This study will give participants the drug for a longer period of time to see if doing this will extend the cancer remission. Clofarabine has been approved by the FDA for the treatment of acute lymphoblastic leukemia (ALL), another form of acute leukemia. The study drug is considered experimental for AML because it has not been approved by the Food and Drug Administration (FDA) for the treatment of AML.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute myeloid leukemia, in first or second remission.
* Age 55 or older
* Patients must have given signed, informed consent prior to registration on study.
* Participants must have attained a complete remission (CR) to induction chemotherapy and are not good candidates for further intensive chemotherapy or a transplant.
* Female patients of childbearing potential must have a negative serum pregnancy test within 2 weeks prior to enrollment.
* Male and female patients must use an effective contraceptive method during the study and for a minimum of 6 months after study treatment.

Exclusion Criteria:

* Patients with a diagnosis of acute promyelocytic leukemia are not eligible.
* Participants cannot be currently receiving chemotherapy, radiation therapy, or immunotherapy.
* Patients must not be receiving any other investigational agents.
* Participants cannot have Hepatitis B or C or HIV.
* Patients must not have an uncontrolled infection

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-06

PRIMARY OUTCOMES:
Determine the maximum tolerated dose of oral clofarabine. | at study completion (estimated at 2 years)

SECONDARY OUTCOMES:
Measure the relapse-free survival. | labs drawn weekly (first cycle) and every other week thereafter until progression

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Altman, MD, Principal Investigator — Northwestern University